CLINICAL TRIAL: NCT01524510
Title: Open, Prospective Study for the Validation of the Predictive Value of Upper Airway Segmentation and CFD Analysis on Outcome Parameters of the Mandibular Replacement Appliance (MRA) Therapy in Obstructive Sleep Apnea Hypopnea Syndrome OSAHS) Patients
Brief Title: Validation of Functional Imaging as Predictive Tool for Outcome of Mandibular Replacement Appliance Therapy in Obstructive Sleep Apnea Hypopnea Syndrome Patients
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: University Hospital, Antwerp (Other)
Responsible Party: Principal Investigator, Wilfried De Backer, Prof. Dr., University Hospital, Antwerp
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: PML_DOC_1101
Record Dates: First submitted 2012-01-23; First posted 2012-02-02 (Estimated); Last update posted 2015-05-28 (Estimated); Status verified 2015-05

CONDITIONS: Obstructive Sleep Apnea Syndrome
Keywords: OSAS; AHI; MRA; CFD
MeSH Terms: conditions — Sleep Apnea, Obstructive

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- MRA (Experimental): All OSAS patients will be asked to sleep two nights without MRA and, +/- 1 week later, two nights with MRA
  Interventions: Radiation: CT scan; Device: Alice PDx polygraphy

INTERVENTIONS:
Radiation: CT scan — low dose radiation scan without contrast without and with MRA
Device: Alice PDx polygraphy — Alice PDx polygraphy (Respironics)

SUMMARY:
In this open prospective study 40 patients who received Mandibular Replacement Appliance (MRA) Therapy as treatment of Obstructive Sleep Apnea Hypopnea Syndrome (OSAHS) will be included. The patient's sleep will be registered during 2 periods of 2 days: one while the patient does not wear the MRA and, +/- 1 week later, one while the patient wears the MRA. Furthermore, 2 low dose CT scans (one with and one without the MRA device in the mouth) will be taken. These data must allow the investigators to validate the use of functional imaging (segmentation and Computational Fluid Dynamics) as a predictor of the outcome of the MRA therapy in OSAHS patients.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with documented OSAHS based on the following criteria:

   AHI >= 5 Complaints of extreme daytime sleepiness with no other explanation and/or 2 or more of the following symptoms:
   * choking or gasping during sleep
   * recurrent awakenings from sleep
   * un-refreshing sleep
   * daytime fatigue
   * impaired concentration
2. Patients who received MRA as treatment for OSAHS
3. AHI >= 5 on at least 1 of the screening nights (patient does not wear MRA device)
4. Male or female patients aged ≥ 18 years
5. Patients with a co-operative attitude
6. Written informed consent obtained

Exclusion Criteria:

1. Pregnant or lactating females or females at risk of pregnancy
2. Patients with an uncontrolled disease or any condition that might, in the judgement of the investigator, place the patient at undue risk or potentially compromise the results or interpretation of the study.
3. Cancer or any other chronic disease with poor prognosis and/or affecting patient status
4. History of alcohol or drug abuse in the last 2 years
5. Patients unlikely to comply with the protocol or unable to understand the nature, scope and possible consequences of the study
6. Patients who participate in another clinical study whose investigational plan is judged to interfere or affect any of the measures of this study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2011-02; Primary Completion 2016-04 (Estimated)

PRIMARY OUTCOMES:
changes in mean AHI between visit 1 and visit 2 | visit 1 (AHI of 2 nights without MRA) / visit 2 (AHI of 2 nights with MRA) (visit 2 happens +/- 1 week after visit 1)
  evaluate the predictive value of upper airway segmentation and CFD analysis on responsiveness to MRA therapy in OSAHS patients
changes in UA resistance | 1 CT scan without MRA (UA resistance without MRA) / 1 CT scan with MRA (UA resistance with MRA)
  evaluate the predictive value of upper airway segmentation and CFD analysis on responsiveness to MRA therapy in OSAHS patients

SECONDARY OUTCOMES:
changes in mean ESS between visit 1 and visit 2 | visit 1 (ESS of 2 nights without MRA) / visit 2 (ESS of 2 nights with MRA) (visit 2 happens +/- 1 week after visit 1)
  to assess the effect of the MRA therapy on daytime sleepiness with the Epworth Sleepiness Scale (ESS).

CONTACTS AND LOCATIONS:
Locations (1):
- UZA, Edegem, Antwerp, Belgium